CLINICAL TRIAL: NCT02769130
Title: Pilot Trial: the Safety and Feasibility of Losartan Therapy for Treatment of Pulmonary Vein Stenosis in Pediatric Patients
Brief Title: Pilot Trial: the Safety and Feasibility of Losartan for Pulmonary Vein Stenosis
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to Health Canada losartan recall, a new formulation being added to the protocol/ temporary suspension
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Christopher Caldarone, Surgeon in Chief, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000051475
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Vein Stenosis; Children
MeSH Terms: conditions — Stenosis, Pulmonary Vein | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Losartan (Experimental): Losartan will be given to children with stenosis in greater or equal to 2 pulmonary veins.
  Maintenance daily dosing is 1mg/kg/day using suspension or tablet formulation of losartan. Losartan will be given for 1 year.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Losartan is given for 12 months
  Other Names: Cozaar

SUMMARY:
This pilot study evaluates the safety and feasibility of losartan in pediatric patients with pulmonary vein stenosis.

It is an open label single arm interventional study. The patient population involves pediatric patients with stenosis in 2 or more pulmonary veins. Patients will be given losartan for 1 year. Outcomes include measures of safety/adverse events and progression of pulmonary vein stenosis.

DETAILED DESCRIPTION:
This pilot study evaluates the safety and feasibility of losartan in pediatric patients with pulmonary vein stenosis.

Large animal studies have demonstrated that losartan can ameliorate the progression of pulmonary vein stenosis in a surgical model of pulmonary vein stenosis.

There is no safety data for losartan in children < 6months of age or in children with pulmonary vein stenosis. Therefore, this study will test the safety and feasibility of losartan in children in an open label single arm interventional study.

Patient inclusion criteria includes stenosis involving 2 or more pulmonary veins. Patients who are consented into the trial with be on losartan therapy for one year. They will undergo study visits every 3 months. Patients will be screened for adverse events through biochemical tests, routine clinical tests and questionnaires.

An exploratory efficacy analysis will compare progression of pulmonary vein stenosis in children enrolled in losartan to a contemporary cohort of children with pulmonary vein stenosis, who did not receive losartan.

ELIGIBILITY:
Inclusion Criteria:

* Stenosis involving 2 or more pulmonary veins
* Consent of parent/legal guardian or child(when appropriate)

Exclusion Criteria:

* History of angioedema or allergic reaction to angiotensin converting enzyme inhibitors
* corrected gestational age of less than 40 weeks
* severe renal dysfunction
* pregnancy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Safety:Number of participants with adverse events | 12 months
  adverse events include hypotension, hyperkalemia, renal dysfunction
Feasibility:Number of participants eligible and recruited | 12 months
  includes patient recruitment and compliance with protocol

SECONDARY OUTCOMES:
Progression of pulmonary vein stenosis: survival | 12 months
  Progression of pulmonary vein stenosis measures include survival, morbidity and evidence of progression on clinical tests

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Caldarone, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No